CLINICAL TRIAL: NCT03790059
Title: Radiofrequency Ablation Combined With Local Injection of Recombinant Human Adenovirus Type 5 in the Treatment of Hepatocellular Carcinoma:A Multicenter Prospective Randomized Controlled Trial.
Brief Title: Radiofrequency Ablation Combined With Recombinant Human Adenovirus Type 5 in the Treatment of Hepatocellular Carcinoma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, fengkai, Principal Investigator, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWH2016LCYB-11
Record Dates: First submitted 2018-12-23; First posted 2018-12-31 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: radiofrequency ablation; hepatocellular carcinoma; recombinant human adenovirus type 5 injection
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RFA combined with H101 group (Experimental): The experimental group was RFA combined H101.H101 has oncolysis in HCC after RFA and reduce tumor recurrence.
  Interventions: Drug: H101; Procedure: RFA
- Conventional RFA group (Other): The standard control group was the conventional RFA.Using RFA for the treatment of small HCC.The efficacy was compared with that of the experimental group combined with H101.
  Interventions: Procedure: RFA

INTERVENTIONS:
Drug: H101 — Intraoperative injection of H101 can improve the efficacy of RFA in hepatocellular carcinoma.
  Other Names: Recombinant Human Adenovirus Type 5 Injection（H101）.
  Arms: RFA combined with H101 group
Procedure: RFA — Treat the samll HCC with the RFA.
  Other Names: Radiofrequency ablation（RFA）.

SUMMARY:
The primary reason for recurrence of hepatocellular carcinoma after radiofrequency ablation (RFA) is the micro-metastatic lesion that has not been ablated and inactivated in the transitional area.Some clinical trials have confirmed that H101(recombinant human adenovirus type 5 injection) has selective oncolysis in a variety of solid tumors.However, there are no reports that H101 which is injected during surgery can improve the efficacy of RFA in liver cancer at present.Therefore,We used a multicenter prospective randomized controlled study as the main method to prospectively compare the short-term and long-term efficacy of RFA combined with H101 group and traditional RFA group in the treatment of small liver cancer (single lesion , diameter less than or equal to 3cm，to evaluate the value of RFA combined with H101 injection in reducing the postoperative recurrence rate of small hepatocellular carcinoma, and to provide a reliable evidence-based medical basis for the selection of treatment methods for small hepatocellular carcinoma.

DETAILED DESCRIPTION:
The primary reason for recurrence of hepatocellular carcinoma after radiofrequency ablation (RFA) is the micro-metastatic lesion that has not been ablated and inactivated in the transitional area.Oncolytic virus H101 is a genetically engineered adenovirus that lacks Elb 55ku protein.Some clinical trials have confirmed that H101 has selective oncolysis in a variety of solid tumors.Furthermore,research shows that the directly dissolving tumor activity of H101 enhanced obviously and activate the body's anti-tumor immune to induce the distal antitumor effect under the condition of mild high temperature (40 ℃ and 42 ℃).The transition zone of RFA can provide the appropriate mild high temperature.However, there are no reports that H101 which is injected during surgery can improve the efficacy of RFA in liver cancer at present.Therefore,We used a multicenter prospective randomized controlled study as the main method to prospectively compare the short-term and long-term efficacy of RFA combined with H101 group and traditional RFA group in the treatment of small liver cancer (single lesion , diameter less than or equal to 3cm，to evaluate the value of RFA combined with H101 injection in reducing the postoperative recurrence rate of small hepatocellular carcinoma, and to provide a reliable evidence-based medical basis for the selection of treatment methods for small hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. The patients understand the content and significance of the study and we obtain a written informed consent from them.
2. The patients' gender are not limited and are between the ages of 18 and 75.
3. Liver function of Child-Pugh Class A or B;The retention rate of indocyanine green for 15 minutes is less than or equal to 20%.
4. The ECOG score is 0.
5. The diagnosis was a single hepatocellular carcinoma with a diameter of no more than 3cm.
6. There were no other related diseases affecting RFA treatment.

Exclusion Criteria:

1. There are tumor emboli in the large vessels of the liver;distant metastasis of HCC.
2. The patient has or has had a history of refractory ascites,hepatic encephalopathy, or esophageal varices hemorrhage.
3. The patient was complicated with other malignant tumors.
4. The patient has severe cardiac, renal and other organ dysfunction.
5. In addition to viral hepatitis, there are other active infectious diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Tumor-free survival | two-years tumor-free survival.
  Postoperative tumor-free survival is an evaluation of tumor recurrence and metastasis.It's also an evaluation of the efficacy of the experimental group

SECONDARY OUTCOMES:
Overall survival | two-years overall survival.
  The percentage of patients who receive certain treatments and are still alive after years of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kuansheng Ma, Ph.D, Study Director — Institute of hepatobiliary surgery,Southwest Hospital
Locations (2):
- China (2):
  - Institute of hepatobiliary surgery,Southwest Hospital, Chongqing, Chongqing Municipality
  - Institute of hepatobiliary surgery,Southwest Hospital, Chongqing